CLINICAL TRIAL: NCT00012792
Title: Randomized Controlled Trial of Exercise Training in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: IIR 96-015
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-12

CONDITIONS: Lung Diseases; Obstructive
MeSH Terms: conditions — Lung Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Exercise Training

INTERVENTIONS:
Behavioral: Exercise Training

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the most common chronic illnesses in the adult population and accounts for approximately 25,000 discharges from VA hospitals in a calendar year. In addition to the burden put on the health care system, COPD is a disabling condition that adversely affects functional status and quality of life (QOL). Several reports have suggested that exercise training programs can reduce the frequency of hospitalization for COPD; however, these reports have important methodological limitations and such programs have not been widely implemented in the VA health care system. Although the underlying lung pathology of COPD may be unalterable, physical reconditioning has been clearly demonstrated to improve cardiorespiratory status in COPD patients. These physiologic changes have the potential to substantially improve QOL and reduce functional disability. Moreover, improved cardiorespiratory reserve may decrease the utilization of health care resources during mild to moderate exacerbation of COPD.

DETAILED DESCRIPTION:
Background:

Chronic obstructive pulmonary disease (COPD) is one of the most common chronic illnesses in the adult population and accounts for approximately 25,000 discharges from VA hospitals in a calendar year. In addition to the burden put on the health care system, COPD is a disabling condition that adversely affects functional status and quality of life (QOL). Several reports have suggested that exercise training programs can reduce the frequency of hospitalization for COPD; however, these reports have important methodological limitations and such programs have not been widely implemented in the VA health care system. Although the underlying lung pathology of COPD may be unalterable, physical reconditioning has been clearly demonstrated to improve cardiorespiratory status in COPD patients. These physiologic changes have the potential to substantially improve QOL and reduce functional disability. Moreover, improved cardiorespiratory reserve may decrease the utilization of health care resources during mild to moderate exacerbation of COPD.

Objectives:

The overall goal of this project is to determine whether exercise training leads to a reduction in chronic institutionalization, acute hospitalization, and outpatient physician visits and to improved functional status and QOL in patients with COPD. The following specific objectives will be accomplished: 1) test the hypothesis that the addition of exercise training to usual care reduces use of health care services over a one-year follow-up period; and 2) test the hypothesis that exercise training leads to improvements in functional status and QOL.

Methods:

Hypotheses will be tested by means of a randomized controlled trial involving subjects with COPD (aged 50-79 years) who receive care at two Boston area VA hospitals. Subjects randomized to the intervention group receive an eight-week program of thrice-weekly exercise training sessions. Outcomes include a standardized QOL questionnaire and objective tests of functional status (6-minute walk and activities of daily living performance).

Status:

Subject recruitment and interventions completed; data collection completed; currently analyzing data on effects of intervention on health care utilization and other parameters.

ELIGIBILITY:
Inclusion Criteria:

COPD diagnosis; FEV,<_ 60% pred; FEV, /FVC< _85% pred

Exclusion Criteria:

Ages: 50 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David William Sparrow, DSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States